CLINICAL TRIAL: NCT02496273
Title: Phase 1 Study of CEA Specific Cytotoxic T Lymphocytes Induced by Dendritic Cells Infected by Recombinant Adeno-associated Virus With CEA Gene in Stage IV Gastric Cancer
Brief Title: Phase I Trial of CEA Specific AAV-DC-CTL Treatment in Stage IV Gastric Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZYY-CTL-001
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Gastric Cancer
Keywords: Dendritic Cells; Cytotoxic T-Lymphocytes; Adeno-Associated Virus
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CEA Specific CTL (Experimental): Patients receiving CEA-specific CTLs as therapy for Gastric Cancer
  Interventions: Biological: CTL

INTERVENTIONS:
Biological: CTL — Mononuclear cells (Dendritic Cell,DC precursor) were isolated from the peripheral blood of gasric cancer by density gradient centrifugation and infected with rAAV/CEA virus.Maturation of the DC was induced by granulocyte-macrophage colony-stimulating factor (GM-CSF), interleukin-4 (IL-4) and tumor necrosis factor-alpha(TNF-alpha). On day 7, the DCs were collected and mixed with T cells at the ratio of 1 to 20 to induce cytotoxic T lymphocytes (CTL).The cells will be proliferated and infused by intravenous (IV) infusion into the patient.
  Other Names: CEA Specific Cytotoxic T-Lymphocytes

SUMMARY:
The purpose of this study is to evaluate the clinical safety and preliminary efficacy of CEA specific cytotoxic T lymphocytes induced by dendritic cells infected by recombinant adeno-associated virus with CEA gene in the treatment of stage IV gastric cancer patients.

DETAILED DESCRIPTION:
Carcinoembryonic antigen (CEA) describes a set of highly related glycoproteins involved in cell adhesion.CEA is normally produced in gastrointestinal tissue during fetal development, but the production stops before birth. The serum levels are raised in some types of cancer,such as Gastric Cancer.The expression of CEA in these cancers and succedent unfavourable prognosis such as tumor hyperplasia, recurrence make CEA become the desirable therapeutic target.

Cancer immunotherapy is the use of the immune system to treat cancer. Immunotherapies fall into three main groups: cellular, antibody and cytokine.Cellular therapies involve the removal of immune cells from the blood or from a tumor. Immune cells specific for the tumor are activated, cultured and returned to the patient where the immune cells attack the cancer. Cytotoxic T cells and dendritic cells can be used in cell-based immunotherapy.

This study is for patients that have a stage Ⅳ gastric cancer with elevated serum CEA concentration. This research study uses special immune system cells called CEA-specific cytotoxic T lymphocytes , a new experimental therapy.

Blood will be collected from the patient and the CEA-specific CTLs will be made.The cells will be injected by IV into the patient.The investigators will follow the patient from their last infusion,monitor side effects of immunotherapy and learn more about the way the T cells are working in the patient's body.The investigators will use blood samples to see how long the T cells last and to look at the immune response to the patient's response to cancer.

ELIGIBILITY:
Inclusion Criteria:

* Any patient, at least 18 yrs old regardless of sex, with a diagnosis of Stage IV Gastric Cancer
* Patients with life expectancy greater than or equal to 6 weeks.
* Patients with a Karnofsky score of greater than or equal to 80.
* serum CEA ≥ 20ng/ml.
* Patient provides consent for all required biopsies.

Exclusion Criteria:

* Patients with severe active infection.
* Patients receiving systemic corticosteroid within 48 hours of CTL infusion.
* Patients with HBV,HCV,HIV infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
ELISPOT assays | 1 month
  Enzyme-Linked ImmunoSpot (ELISPOT) assay is used for monitoring CEA specific cellular immune responses in Gastric Cancer

SECONDARY OUTCOMES:
overall survival (OS) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Wu Changping, M.D, Study Chair — The First People's Hospital of Changzhou

REFERENCES:
- [Background] Caruana I, Weber G, Ballard BC, Wood MS, Savoldo B, Dotti G. K562-Derived Whole-Cell Vaccine Enhances Antitumor Responses of CAR-Redirected Virus-Specific Cytotoxic T Lymphocytes In Vivo. Clin Cancer Res. 2015 Jul 1;21(13):2952-62. doi: 10.1158/1078-0432.CCR-14-2998. Epub 2015 Feb 17. PMID 25691731
- [Background] Cui H, Zhang W, Hu W, Liu K, Wang T, Ma N, Liu X, Liu Y, Jiang Y. Recombinant mammaglobin A adenovirus-infected dendritic cells induce mammaglobin A-specific CD8+ cytotoxic T lymphocytes against breast cancer cells in vitro. PLoS One. 2013 May 1;8(5):e63055. doi: 10.1371/journal.pone.0063055. Print 2013. PMID 23650543
- [Background] Martino AT, Basner-Tschakarjan E, Markusic DM, Finn JD, Hinderer C, Zhou S, Ostrov DA, Srivastava A, Ertl HC, Terhorst C, High KA, Mingozzi F, Herzog RW. Engineered AAV vector minimizes in vivo targeting of transduced hepatocytes by capsid-specific CD8+ T cells. Blood. 2013 Mar 21;121(12):2224-33. doi: 10.1182/blood-2012-10-460733. Epub 2013 Jan 16. PMID 23325831